CLINICAL TRIAL: NCT03734224
Title: Inguinal Hernia Operation and Postoperative Pain - a Prospective and Randomized Study
Brief Title: Inguinal Hernia Operation and Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anna-Maria Thölix, MD, Surgical resident, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS-459-2018-61
Record Dates: First submitted 2018-10-27; First posted 2018-11-07 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Pain, Postoperative; Inguinal Hernia; Quality of Life
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1: Adhesix (Active Comparator): This group gets the Adhesix mesh in a normal open hernia operation.
  Interventions: Procedure: Adhesix mesh
- Group 2: Progrip (Active Comparator): This group gets the Progrip mesh in a normal open hernia operation.
  Interventions: Procedure: Progrip mesh

INTERVENTIONS:
Procedure: Adhesix mesh — Adhesix mesh
  Arms: Group1: Adhesix
Procedure: Progrip mesh — Progrip mesh
  Arms: Group 2: Progrip

SUMMARY:
Inguinal hernia is a common disease, which is treated surgically when symptomatic. Pain after open inguinal hernia surgery can affect the patient significantly and weaken their quality of life. The aim of this study is to find out if the choice of mesh affects postoperative pain and therefore causes more contacts to the health care center. Our goal is also to find out how the pain affects the patients´ quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old male patients, with a symptomatic inguinal hernia that can be diagnosed by clinical examination. Primary and unilateral hernia. The operation performed at a day surgery unit.

Exclusion Criteria:

* female
* bilateral hernia
* Incarcerated hernia
* Scrotal hernia
* ASA-classification >3
* BMI >35 or <18
* No hernia found in clinical examination
* Liver cirrhosis
* Other contraindication for inguinal hernia operation
* Anticoagulant therapy, that needs bridge therapy when paused

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of contacts due to postoperative pain | 3 months
  Number of postoperative contacts to the operating unit due to pain at 3 months after the operation

SECONDARY OUTCOMES:
The use of pain medication | 1 year
  The use of painkillers postoperatively
Pain intensity | 1 year
  The pain intensity at the Numeric Pain Rating Scale (NPRS), where the 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine")
Number of contacts | 1 year
  Number of contacts to the operating unit/health care system due to pain after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University hospital, Jorvi hospital, Espoo, Finland

REFERENCES:
- [Derived] Tholix AM, Kossi J, Harju J. One-year outcome after open inguinal hernia repair with self-fixated mesh: a randomized controlled trial. Langenbecks Arch Surg. 2023 Sep 21;408(1):369. doi: 10.1007/s00423-023-03106-w. PMID 37733083